CLINICAL TRIAL: NCT02459405
Title: Decreasing Leak Rate in Colorectal Surgery Using Near Infra-red (NIR) Imaging: a Multicentric Prospective Phase II Study
Brief Title: Decreasing Leak Rate in Colorectal Surgery Using Near Infra-red (NIR) Imaging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); University College Dublin (Other)
Responsible Party: Principal Investigator, Ris Frederic, MD, PD, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10/H0724/13
Record Dates: First submitted 2015-04-04; First posted 2015-06-02 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Anastomotic Leak
Keywords: Colorectal surgery; Near infrared; Indocyanine green; anastomotic leak; Prevention of leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIR anastomotic perfusion assessment (Experimental): Patient will have their anastomosis assessed after they receive 7.5 to 9 mg of Indocyanine green intravenously (at a concentration of 2.5mg/ml).
  The microvascularisation assessment will be performed using a near infrared device(Pinpoint device), allowing to increase reality.
  This procedure will be repeated twice during the surgery, the first time before and the second time after the anastomosis has been done.
  Interventions: Procedure: NIR anastomotic perfusion assessment; Device: Near infrared camera

INTERVENTIONS:
Procedure: NIR anastomotic perfusion assessment — Patient will have their anastomosis assessed by near infrared technology after indocyanine green has been injected i.v. The procedure will be repeated twice, once before the anastomosis and the second time after the anastomosis has been performed.
  Other Names: Indocyanine assessment of anastomotic microvascularisation
Device: Near infrared camera — Use of the Pinpoint laparoscopic scope (Novadaq, Vancouver, Canada) after injection of indocyanine green
  Other Names: Pinpoint evaluation

SUMMARY:
Anastomotic leak is a devastating complication of colorectal surgery. There is no widespread means of assessing the viability of a laparoscopic anastomosis. The investigators described recently the feasibility of microvascularisation assessment with near-infra red technology (NIR).

The aim of this study is to look at the implementation of this technique in a wider prospective series of patients undergoing colorectal resection.

DETAILED DESCRIPTION:
Multicentric prospective study of 260 consecutive patients undergoing colonic resection and being assessed during the course of surgery for microvascularisation.

After vessel division and after colorectal anastomosis, indocyanine green (2.5mg/ml) is injected intravenously and anastomotic microvascularisation assessed with the PinPoint NIR system (Novadaq, Vancouver, Canada).

Study primary endpoint is the anastomotic leak rate Secondary endpoint are peroperative and post-operative complications according to the Clavien Dindo scale, time of the procedure and time to record a signal as well as any change of the procedure.

This study will be performed on 3 different sites Geneva, Oxford and Dublin University Hospitals

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Participant willing and able to comply with the study procedures.
* Diagnosed with required colon or rectal neoplasia requiring surgical excision by either laparoscopic or open surgery.
* A negative pregnancy test for women of childbearing potential prior to surgery
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Allergy to Indocyanine green.
* Participant who is undergoing purely palliative surgery or who is terminally ill
* Subject has other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2013-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak rate | first 30 days
  anastomotic leak rate at 30 post operative days

SECONDARY OUTCOMES:
Time to perform the near infrared procedure | during surgery
  measured added time to the procedure
Time to get a near infrared signal | during surgery
  Time to see a signal during surgery
complication rate | 30 days
  according to Clavien Dindo classification
Mortality | 30 days
  30 days mortality
Alteration of the course of surgery due to insufficient vascularisation | during surgery
  If the vascularisation is insufficient during the surgery, the investigators can change the course of the surgery he is performing. For example, it could lead to a second resection to obtain well vascularized tissue for the anastomosis. Any alteration of the regular course of surgery for the safety of the patient is reported. The number of patient requiring an alteration of the course of surgery will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Ris, MD, Prof, Principal Investigator — University Hospital, Geneva
Locations (4):
- Dublin University College, department of colorectal surgery, Dublin, Ireland
- Humanitas Universtity Hospitals, Milan, Rozzano (Milano), Italy
- Geneva University Hospitals, Service of Visceral Surgery, Geneva, Switzerland
- Oxford University Hospitals, Department of colorectal Surgery, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Ris F, Hompes R, Cunningham C, Lindsey I, Guy R, Jones O, George B, Cahill RA, Mortensen NJ. Near-infrared (NIR) perfusion angiography in minimally invasive colorectal surgery. Surg Endosc. 2014 Jul;28(7):2221-6. doi: 10.1007/s00464-014-3432-y. Epub 2014 Feb 25. PMID 24566744
- [Background] Cahill RA, Ris F, Mortensen NJ. Near-infrared laparoscopy for real-time intra-operative arterial and lymphatic perfusion imaging. Colorectal Dis. 2011 Nov;13 Suppl 7:12-7. doi: 10.1111/j.1463-1318.2011.02772.x. PMID 22098511
- [Derived] Ris F, Liot E, Buchs NC, Kraus R, Ismael G, Belfontali V, Douissard J, Cunningham C, Lindsey I, Guy R, Jones O, George B, Morel P, Mortensen NJ, Hompes R, Cahill RA; Near-Infrared Anastomotic Perfusion Assessment Network VOIR. Multicentre phase II trial of near-infrared imaging in elective colorectal surgery. Br J Surg. 2018 Sep;105(10):1359-1367. doi: 10.1002/bjs.10844. Epub 2018 Apr 16. PMID 29663330